CLINICAL TRIAL: NCT04682470
Title: COMPRehensive Assessment of Prevalence, Risk Factors and Mechanisms of Impaired Medical and Psychosocial Health Outcomes Among Adolescents and Young Adults With Cancer: the Prospective Observational COMPRAYA Cohort Study
Brief Title: The Prospective Observational COMPRAYA Cohort Study
Acronym: COMPRAYA
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: M20COM
Record Dates: First submitted 2020-11-16; First posted 2020-12-23 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Second Cancer; Survivorship; Fertility Issues; Distress, Emotional; Lifestyle; Genetic Disease; Cancer
MeSH Terms: conditions — Neoplasms, Second Primary; Infertility; Genetic Diseases, Inborn; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Other: No intervention ; observational

INTERVENTIONS:
Other: No intervention ; observational — No intervention; observational

SUMMARY:
Rationale: Childhood cancer survivorship attracts attention globally, because successes in treatment have led to increasing number of survivors who reach adulthood, in which survivorship issues affecting health-related quality of life (HRQoL) become prominent. Most paediatric patients are treated intensively with irradiation and/or chemotherapy, which put them at risk for early and/or late adverse medical and psychosocial events. In contrast, much less is known about adolescent and young adult (AYA) cancer patients, diagnosed between 18-39 years, who, with an 80% chance to survive, also have a long life ahead. AYA cancer patients, much more than children, suffer from delay in diagnosis, lack of centralization of care, ageadjusted expertise, and AYA follow-up care. AYAs typically present with a rare tumour: either with a paediatric malignancy (e.g. acute lymphoblastic leukaemia, paediatric brain tumours), a more typical tumour of AYA age (e.g. Hodgkin's disease, germ cell cancer, melanoma, thyroid cancer) or with an adult tumour at unusual young age (e.g. gastrointestinal, lung, breast carcinomas). Next to these differences in epidemiology, the tumour biology, developmental challenges (e.g. forming relationships, becoming financially independent, having children) and treatment regimens differ between AYAs and children, and therefore findings derived from childhood cancer survivors cannot be extrapolated to AYAs. Furthermore, novel treatments with targeted agents or immunotherapy are more likely to be administrated to AYAs compared to children. Finally, a rare group of incurable AYA cancer patients will survive for many years, for whom health outcome and supportive care intervention data are lacking.

Globally, so far, the identification of AYA cancer patient subgroups that might be more susceptible to poor health outcomes has not been systematically addressed. The role of sociodemographic and treatment-associated risks, external exposures (e.g. lifestyle) and host factors (e.g. genetic, biological, physiological); or combinations of influences for impaired (agespecific) health outcomes, remains largely unknown. Understanding who is at risk and why will support the development of evidence-based AYA prevention, treatment and supportive care programs and guidelines, in co-creation with AYA cancer patients.

Objective: To examine the prevalence, risk factors and mechanisms of impaired health outcomes (short- and long-term medical and psychosocial effects and late effects) over time among a population-based sample of AYA cancer patients.

Study design: Prospective, observational cohort study Study population: All AYAs diagnosed (18-39 years at primary diagnosis) with cancer (any type) within the first 3 months after diagnosis (eligibility window of 1 month to ensure all eligible AYA cancer patients can be included) in one of the participating centres (or treated in one of these centres) in The Netherlands.

Main study parameters/endpoints: The main outcomes are medical (e.g. second tumour; survival; fertility) and psychosocial (e.g. distress) health outcomes. Other study parameters (covariates/moderators/mediators) are characteristics of the individual (e.g. age, sex, cultural background, partner status, educational level, occupation, tumour type, disease stage, body composition, comorbid conditions, coping style), characteristics of the environment (e.g. cancer treatment, lifestyle), and genetic and biological factors (e.g. family history of cancer, stress and inflammation markers (e.g. cortisol, IL-6), microbiome).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: On an individual level, patients who participate are asked to complete questionnaires on an annual basis for at least 10 years. All sample collections will take place at three time points: 0-3 months after diagnosis (baseline), 2 and 5 years; except blood for DNA analyses which will only take place at baseline. The collection of blood, hair and faeces at three occasions is minimally invasive and the risks of blood draws, hair and fecal sampling are negligible. All safety measures and procedures will be performed according to local guidelines. Patients will not experience direct benefit from participation in the COMPRAYA study.

By participating, patients will contribute to a better insight in the prevalence of impaired medical and psychosocial (age-specific) health outcomes in AYA and evidence on factors associated with these health outcomes. This will lead to better and more personalized cancer care and supportive care tools for future AYA cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed cancer diagnosis;
* Age 18 - 39 years at time of first cancer diagnosis;
* Able to understand the informed consent form;
* Provide written informed consent.

Exclusion Criteria:

* Mentally incompetent patients based on the opinion of treating physician .
* Inability to understand the Dutch language
* Life expectancy less than 6 months based on the opinion of treating physician .

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All AYA cancer patients, diagnosed at age 18-39 years in one of the participating hospitals,receive an invite within the first 3 months after diagnosis (eligibility window of 1 month to ensure all eligible AYA cancer patients can be included) and will be asked to complete the COMPRAYA questionnaires on an annual basis up to 10 years after diagnosis (again with a window of 2 months before and after). Collection of clinical data and samples (e.g. faeces, hair and blood) will be done at baseline, 2, and 5 years after diagnosis. Questionnaire data collection is guaranteed by the PROFILES registry and patients will give informed consent for linkage with registry data, which makes long-term follow-up possible.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Second tumor | Change from baseline throughout follow-up of 10 years
  Linkage to the Netherlands Cancer Registry (NCR) to asses second malignancies.
Survival | Change from baseline throughout follow-up of 10 years
  Linkage will done with the Personal Records Database (BRP) to have information on survival status.
Distress | Change from baseline throughout follow-up of 10 years
  Psychological distress will be assessed at each time point with the Hospital Anxiety and Depression Scale (HADS), with seven items each for assessing symptoms of anxiety and depression. Answers range from 0 to 3 and scores for each subscale are calculated by addition of the items, with a higher score meaning more anxiety or depression.
Fertility problems and wish for children | Change from baseline throughout follow-up of 10 years
  A questionnaire will be used to asses fertility problems and their wish for children. Linkage will be done to the Netherlands Perinatal Registry (NPR) to receive data about pregnancy and children.
Health related quality of life | Change from baseline throughout follow-up of 10 years)
  The EORTC QLQ-C30 is a 30-item HRQoL questionnaire consisting of five functional scales (physical, role, cognitive, emotional and social), a global quality of life scales, symptom scales (fatigue, pain, nausea and vomiting) and a number of single items assessing common symptoms (dyspnea, loss of appetite, sleep disturbance, constipation and diarrhea) and perceived financial impact of the disease. After linear transformation, all scales and single item measures range in score from 0-100. A higher score on the functional scales and global QoL means better functioning and HRQoL, whereas a higher score on the symptom scales means more complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Husson, Phd, Principal Investigator — Netherlands Cancer Institute- Antoni van Leeuwenhoek Hospital (NKI-AvL); Winette van de Graaf, Prof, Study Director — Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital (NKI-AvL)
Locations (1):
- Antoni van Leeuwenhoekziekenhuis, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT04682470/Prot_SAP_000.pdf